CLINICAL TRIAL: NCT06290596
Title: Vasopressin Versus Tranexamic Acid for Control of Blood Loss Related to Abdominal Hysterectomy: A Randomized Clinical Study
Brief Title: Vasopressin Versus Tranexamic Acid for Control of Blood Loss Related to Abdominal Hysterectomy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Warda Demerdash Khalifa Ali, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSR/AZAST/AIP029/21/222/8/2023
Record Dates: First submitted 2024-02-27; First posted 2024-03-04 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Uterine Surgery
MeSH Terms: interventions — Vasopressins; Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vasopressin group (Experimental): patients in this group will be injected with a 10-ml syringe containing 10 units of vasopressin (5 mL bilaterally)
  Interventions: Drug: Vasopressin
- Tranexamic acid group (Experimental): patients in this group will be injected with a 10-ml syringe containing 10 ml of tranexamic acid (5 mL bilaterally).
  Interventions: Drug: Tranexamic acid
- Control group (Placebo Comparator): patients in this group will be injected with a 10-ml syringe containing 10 ml of normal saline (5 mL bilaterally).
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Vasopressin — Hemostatic drug.
  Arms: Vasopressin group
Drug: Tranexamic acid — Hemostatic drug.
  Arms: Tranexamic acid group
Other: Saline — Placebo
  Arms: Control group

SUMMARY:
To find the best option to reduce blood loss related to abdominal hysterectomy (AH), the present randomized double-blinded study sought to compare the effects of locally administered vasopressin (VP) and tranexamic acid (TXA) on blood loss in women submitted to AH for benign lesions.

DETAILED DESCRIPTION:
To find the best option to reduce blood loss related to abdominal hysterectomy (AH), the present randomized double-blinded study sought to compare the effects of locally administered vasopressin (VP) and tranexamic acid (TXA) on blood loss in women submitted to AH for benign lesions.

Interventions Study interventions Patients in all groups will receive identically looking pharmaceutical preparations which differ according to the study group

1. Vasopressin group Just before beginning of AH, patients in this group will be injected with a 10-ml syringe containing 10 units of VP (5 mL bilaterally), 1 cm medial to the uterine vessels in the most distal area of the lower uterine segment not to compromise the bladder. If this site is not accessible, patients will be alternatively injected in the midline at the fundus (Okin et al., 2001). In addition, and just before closure of peritoneum, 100 ml of normal saline (NS) will be applied topically over the raw surface.
2. Tranexamic acid group Just before AH, patients in this group will be injected with a 10-ml syringe containing 10 ml of NS (5 mL bilaterally) as described above. Just before closure of peritoneum, 1.5 g of TXA mixed in 100 ml of NS will be applied topically over the raw surface (Mitra et al., 2022).
3. Control group Just before AH, patients in this group will be injected with a 10-ml syringe containing 10 ml of NS (5 mL bilaterally) as described above. In addition, and just before closure of peritoneum, 100 ml of normal saline (NS) will be applied topically over the raw surface.

ELIGIBILITY:
Inclusion Criteria:

- Patients will be included in the present study if they are indicated for abdominal hysterectomy for benign lesions.

Exclusion Criteria:

* history of coagulation or bleeding disorders or
* if they were under antithrombotic treatment.
* associated malignancy, renal impairment or allergy to TA.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 387 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
blood loss | 24 hours
  Amount of blood loss in mL

IPD SHARING:
Plan to Share IPD: No